CLINICAL TRIAL: NCT00931424
Title: The Clinical Research of Surgery on Primary Chronic Venous Insufficiency
Brief Title: The Clinical Trial for Primary Chronic Venous Insufficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: wang shen-ming, The first affiliated hospital of Sun Yat-Sen university
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008001
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-05

CONDITIONS: Primary Chronic Venous Insufficiency
Keywords: Primary Chronic Venous Insufficiency; surgery; reconstruction; valve

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- reconstruction (Experimental): patients in this group will have both valve reconstruction and superficial vein surgery
  Interventions: Procedure: valve reconstruction
- unreconstruction (No Intervention): patients in this group will only have superficial vein surgery

INTERVENTIONS:
Procedure: valve reconstruction — reconstruct valve at the same time of superficial vein surgery
  Arms: reconstruction

SUMMARY:
A multicenter Random Clinical Trial to confirm the advantage of the valve reconstructive surgery on Primary Chronic Venous Insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* PCVI patients with III degree back flow in deep vein that is confirmed by color doppler or phlebography

Exclusion Criteria:

* age over 70 years old
* pregnancy
* patients with severity arteriosclerosis obliterans, malignancy, severity disease of heart, lung or brain, and hematopathy

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
clinical-etiology-anatomic-pathophysiologic classification system | 3 month, 1 year, 3 year, 5 year, 7 year

SECONDARY OUTCOMES:
phlebography | 3 month, 1 year, 3 year, 5 year, 7 year
color doppler | 3 month, 1 year, 3 year, 5 year, 7 year

CONTACTS AND LOCATIONS:
Overall Officials: Shen-ming Wang, doctor, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The first affiliated hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China